CLINICAL TRIAL: NCT02699918
Title: Impact of Obstructive Sleep Apnea Syndrome on Metastatic Potential of Cutaneous Melanoma : Prospective Study in Patients With High Risk Melanoma
Brief Title: Impact of Obstructive SAS on Metastatic Potential of Cutaneous Melanoma
Acronym: MELA-SAS
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: failure in regulatory statements
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Agiradom
Record Dates: First submitted 2015-12-22; First posted 2016-03-07 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Melanoma With a Breslow's Thickness ≥ 1mm; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- screening oxymetry (Experimental): nocturnal oxymetry to screen for sleep apnea
  Interventions: Procedure: nocturnal oximetry

INTERVENTIONS:
Procedure: nocturnal oximetry — nocturnal oximetry for screening of sleep apnea syndrome. Patients with abnormal nocturnal oximetry will be further explored by polysomnography.

SUMMARY:
Hypothesis: to address if diagnosis of obstructive sleep apnea before or during the extending check-up is a risk factor toward metastasis for melanoma stage ≥ tIIaN0M0 Study design: Adult patients with a Breslow's Thickness ≥ 1mm coming to the surgery consultation will have a nocturnal oximetry for screening of obstructive sleep apnea. Patients having an abnormal nocturnal oximetry will be explored by polysomnography in order to detect sleep apnea syndrome. Patients with sleep apnea will be treated.

Standard dermatologic follow-up over a 3 years period with thoraco-abdominal-pelvic and cerebral CT-scan and a lymph-node ultrasound every 6 months will be performed.

DETAILED DESCRIPTION:
Melanoma is a cutaneous cancer due to a proliferation of melanocytes. For metastatic cases the prognostic is poor (18% survival at 5 years). Few factors predict metastasis. Sleep Apnea Syndrome is involved in mechanism of carcinogenesis and aggressiveness markers of malignant cutaneous melanoma.

Hypothesis: to address if diagnosis of obstructive sleep apnea before or during the extending check-up is a risk factor toward metastasis for melanoma stage ≥ tIIaN0M0 Study design: Adult patients with a Breslow's Thickness ≥ 1mm coming to the surgery consultation will have a nocturnal oximetry for screening of obstructive sleep apnea. Patients having an abnormal nocturnal oximetry will be explored by polysomnography in order to detect sleep apnea syndrome. Patients with sleep apnea will be treated.

Standard dermatologic follow-up over a 3 years period with thoraco-abdominal-pelvic and cerebral CT-scan and a lymph-node ultrasound every 6 months will be performed.

Sample size: based on previous data from the investigators showing that 25% of patients with a Breslow's Thickness ≥ 1mm will have node or visceral metastasis. For an alpha threshold of 5% and a study power of 80%, with 5% of dropouts, with the hypothesis that 40% of apnea syndrome patients will metastasis versus 20% in the control group the study should include 83 patients in each group.

Statistical analysis: an intermediate analysis after 80 included patients will be performed. Peto method will be followed, results will be considered significant with a p≤0.001 and the study will be stopped.

Normality of data will be checked by Kurtosis and Skewness tests, variance equality will be tested with the Leven test. The significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* adults hospitalized in the dermatological unit for the initial consult for a melanoma with a Breslow's Thickness ≥ 1mm

Exclusion Criteria:

* pregnant women
* Institutionalized patient
* patients with metastasis in the lymph node or any organ at the time of the first consult
* patients with another neoplasia requiring treatment other than surgery in the last 5 years
* patients with creatinine above 200µmol/ml or clearance below 30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12-01; Primary Completion 2016-04-01 (Estimated); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Ratio of metastasis confirmed by thoraco-abdominal-pelvic or cerebral CT in patients subgroups with or without sleep apnea syndrome | 3 years period
  sleep apnea is defined witn an Apea Hypopnea Index ≥ 5

SECONDARY OUTCOMES:
Ratio of a positive status of the sentinel lymph node confirmed by histological measurements in patients subgroups with or without sleep apnea syndrome | initial care
  sleep apnea is defined witn an Apea Hypopnea Index ≥ 5
In the subgroup of patients with sleep apnea syndrome, ratio of patients with metastatic evolution according to the CPAP treatment adherence | 3 years
  adherence of CPAP ≥ 4h by night or 3h by night

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Pépin, Pr MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No